CLINICAL TRIAL: NCT05184205
Title: Photodynamic Therapy for SARS-CoV-2 Viral Reduction in the Upper Airway in PCR-positive Asymptomatic Individuals.
Brief Title: Photodynamic Therapy for COVID-19 Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondine Biomedical Inc. (Industry)
Collaborators: University of Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SARS_PDT01
Record Dates: First submitted 2021-12-20; First posted 2022-01-11 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Respiratory Infection; SARS-CoV-2 Acute Respiratory Disease
Keywords: SARS-CoV-2; antimicrobial photodynamic therapy (aPDT); COVID-19; viral load; Nasal decolonization
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a single-center open-label study to evaluate antimicrobial photodynamic therapy (PDT) for upper airway decolonization in patients presenting with SARS-CoV-2 positive antigen test with mild or no symptoms of COVID-19.
Who Masked: Participant
Masking Description: The placebo control arm will include the application of saline isotonic solution and the introduction of the PDT device with no powering on. Due to the characteristics of the device, and the need for the investigator to deliberately not switching it on, it is clear that there cannot be a blind scheme in this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention (Experimental): The procedure is initiated by swabbing the Formulation Applicator, pre-saturated with photosensitizer formulation, inside the patient's nares. The operator then connects the Nasal Light Illuminator (NLI) to the Light Source and inserts the NLIs into the patient's nostrils. The Light Source is turned on, and a 4-minute illumination cycle provides two channels of diffused red light (one for each nostril) to activate the applied formulation. Illumination stops automatically upon completion of the 4-minute cycle. The process is then repeated using two new Formulation Applicators to ensure full disinfection coverage.
  Interventions: Device: Nasal Photodisinfection
- Sham Comparator: Control (Sham Comparator): Sham comparator
  Interventions: Device: Sham Comparator: Control

INTERVENTIONS:
Device: Nasal Photodisinfection — The procedure is initiated by swabbing the Formulation Applicator, pre-saturated with photosensitizer formulation, inside the patient's nares. The operator then connects the Nasal Light Illuminator (NLI) to the Light Source and inserts the NLIs into the patient's nostrils. The Light Source is turned on, and a 4-minute illumination cycle provides two channels of diffused red light (one for each nostril) to activate the applied formulation. Illumination stops automatically upon completion of the 4-minute cycle. The process is then repeated using two new Formulation Applicators to ensure full disinfection coverage.
  Arms: Active Intervention
Device: Sham Comparator: Control — Patients who are SARS-CoV-2 positive whose PCR levels are followed but no active intervention will be done. Saline will be used in their nose and the light device will be inserted but not turned on. Patient will be wearing light protecting glasses.
  Arms: Sham Comparator: Control

SUMMARY:
This is a single-center open-label study to evaluate antimicrobial photodynamic therapy (aPDT) for upper airway decolonization in patients presenting with SARS-CoV-2 positive antigen test with mild or no symptoms of COVID-19.

DETAILED DESCRIPTION:
There is a wide variety of people who test positive for SARS-CoV-2. This is directly dependent upon their exposure to the virus, their age and any medical comorbidities that they may have. At this time, it is not possible to predict who will have an adequate immune response to avoid getting COVID-19. Since this remains unpredictable a universal approach to treating SARS-CoV-2 positive patients may be the optimal approach.

The rational for this study design is that in a real world setting numerous patients across a wide variety of conditions will receive testing for SARS-CoV-2 for a variety of reasons. For those who test positive and are asymptomatic or have only mild symptoms, the current standard of care is observation and quarantine. The incubation period can range from 2-14 days with a mean of 5-6 days. Depending upon an individual's original inoculum of virus, comorbidities and other factors they may progress to COVID-19. Preemptive treatment during this time frame may avoid or mitigate COVID-19 disease severity. In certain high-risk individuals attenuating the disease may avoid hospitalization or death, ICU admission and shorten hospital stays.

The nasal disinfection process rapidly and lethally disrupts the microbial cell wall, leaving human tissue unharmed. The topically applied photosensitizer formulation selectively stains bacteria by binding with microbial cell wall components. The red light is absorbed by the photosensitizer molecules, causing electronic state transitions within the photosensitizer. The excited photosensitizer immediately transfers energy to surrounding molecular oxygen, thereby producing reactive oxygen species (ROS) that are responsible for the lethal cell wall disruption.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female ≥ 18 years of age
4. Patient showing a positive test for SARS-CoV-2 with < 26 Ct of an FDA-approved PCR test who is symptomatic or flu-like illness or pneumonia
5. Ability to tolerate an 12-minute non-painful nasal light illumination

Exclusion Criteria:

1. Inability to tolerate insertion of the light illuminator due to oronasal size, shape, or anatomical variants
2. Known allergic reactions to components of the nasal decolonization treatment including methylene blue or chlorhexidine gluconate.
3. COVID-19 illness that is moderate or severe in nature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 viral titer reduction | Immediately following treatment and on days 3, 7, and 14.
  Change from baseline PCR count with testing on days 3, 7 and 14

SECONDARY OUTCOMES:
General safety of nasal photodisinfection | 14 days post treatment
  Observation for any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Josepmaria Argemi, MD, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: No